CLINICAL TRIAL: NCT04648293
Title: Starling Registry Study
Status: Completed | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BXU553561
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Hemodynamic Monitoring
Keywords: Cardiac Index (CI); Stroke Volume (SV); Stroke Volume Index (SVI); Stroke Volume Variation (SVV); Heart Rate (HR); Ventricular Ejection Time (VET); Total Peripheral Resistance (TPR); Total Peripheral Resistance Index (TPRI); Cardiac Power (CP); Cardiac Power Index (CPI); Blood Oxygenation (SPO2); Oxygen Delivery Index (DO2I); Electrical impedance of the chest cavity (Z0); Thoracic Fluid Content (TFC)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Improvement in Hemodynamics: Over the course of a patient's hospitalization, data will be collected on patients from the initiation to completion of hemodynamic monitoring with the Starling monitor in a wide variety of clinical settings, and for different diagnoses. Improvement in hemodynamics is exhibited by an increase in both Cardiac Output and Stroke Volume observed at 12 hour intervals from time of monitoring until completion.
  Interventions: Device: Starling
- No Improvement in Hemodynamics: Over the course of a patient's hospitalization, data will be collected on patients from the initiation to completion of hemodynamic monitoring with the Starling monitor in a wide variety of clinical settings, and for different diagnoses. No Improvement in hemodynamics is exhibited by no increase in both Cardiac Output and Stroke Volume observed at 12 hour intervals from time of monitoring until completion.
  Interventions: Device: Starling

INTERVENTIONS:
Device: Starling — Starling is a portable, non-invasive, cardiac output detector system. The Starling monitor measures the cardiac output by employing electrical bioreactance that measures the electrical characteristics of a volume of tissue and fluid. In the case of cardiac output measurements, the relevant tissue includes the heart and the immediate surrounding volume of the thorax. The relevant fluid is blood. Baxter Healthcare's Starling electrode is a double electrode sensor. Within each sensor, one electrode is used to transmit a high frequency sine wave into the body, while the resulting voltage is measured at the adjacent electrode. Four electrodes are placed at specific areas of the thorax, the impedance to the current flow calculated, and the electrical bioreactance waveform constructed. This information is used to determine cardiac output, and measures and displays associated hemodynamic parameters based on calculations of measurements already incorporated into the Starling device.

SUMMARY:
Hemodynamic optimization of critically ill patients is a goal for clinicians in order to afford the patient the best possible outcomes. Being able to precisely and rapidly determine patient fluid responsiveness provides the bedside physician and nursing staff the information needed to make critical decisions in regards to the patient's fluid status and management of additional fluids and medications.

As fluid management and cardiac output determination are linked to better decision-making and improved outcomes in ICU, the use of a dynamic assessment of fluid responsiveness becomes a key tool for patient management.

This study is designed to collect treatment and outcome data on patients that have undergone hemodynamic monitoring in a wide variety of clinical settings, involving a variety of patient diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 to 95 years of age
* Patient has undergone hemodynamic monitoring with the Starling monitor
* Hemodynamic monitoring was completed no earlier than 2018

Exclusion Criteria:

* None

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who meet the inclusion criteria within an approximate 12-24 months enrollment period will be included in the study. All patients included in this study with available data will be part of the analysis population.
Sampling Method: Probability Sample
Enrollment: 1207 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
30 day in-hospital mortality rate | Day 1 to Day 30
Number of days on vasopressors | Day 1 to Day 30
Volume of treatment fluid administered | Time of monitoring to completion
Number of participants needing mechanical ventilation | Time of monitoring to completion
Lactate level | Time of monitoring to completion
Number of days in Intensive Care Unit (ICU) | Day 1 to Day 30
Number of days in Hospital | Day 1 to Day 30

SECONDARY OUTCOMES:
Number of participants with COVID-19 | Time of monitoring to completion
Number of participants with COVID-19 by treatment type | Time of monitoring to completion
Number of participants with COVID-19 by outcome type | Time of monitoring to completion
Percent of participants that are fluid responsive | Time of monitoring to completion
Number of participants with diastolic dysfunction | Time of monitoring to completion
Percent of participants with fluid responsiveness in diastolic dysfunction | Time of monitoring to completion
Number of participants with device related Non-Serious Adverse Events | Time of monitoring to completion
Number of participants with device related Serious Adverse Events | Time of monitoring to completion

CONTACTS AND LOCATIONS:
Overall Officials: Caio Plopper, MD, Study Director — Baxter Healthcare
Locations (9):
- United States (9):
  - Baxter Investigational Site, Denver, Colorado
  - Baxter Investigational Site, Quincy, Illinois
  - Baxter Investigational Site, Kansas City, Kansas
  - Baxter Investigational Site, St Louis, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Baxter Investigational Site, Camden, New Jersey
  - Baxter Investigational Site, Cleveland, Ohio
  - Baxter Investigational Site, Columbus, Ohio
  - Baxter Investigational SIte, Galveston, Texas

IPD SHARING:
Plan to Share IPD: Undecided